CLINICAL TRIAL: NCT05018754
Title: Treatment of Oral Mucositis Using Platelet Rich Fibrin: a Retrospective Study in Oncological Patients.
Brief Title: Treatment of Oral Mucositis Using Platelet Rich Fibrin TREATMENT OF ORAL MUCOSITIS USING PRF
Status: Completed | Type: Observational
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Francesco Gianfreda, PhD Student, University of Rome Tor Vergata
Other Study IDs: 25071995
Record Dates: First submitted 2021-08-18; First posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Graft Vs Host Disease; Oral Mucositis (Ulcerative); Mesenchymal Stem Cells
Keywords: PRF; Oral Mucositis
MeSH Terms: conditions — Graft vs Host Disease; Stomatitis; Ulcer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Patients affected by oral mucositis (9 RIOM, 6 chemotherapy-related oral mucositis).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: TREATMENT OF ORAL MUCOSITIS USING PLATELET-RICH-FIBRIN (PRF) — All patients were affected by oral mucositis (9 RIOM, 6 chemotherapy-related oral mucositis). They were treated with almost 2 different systemic therapies before and during platelets gel applications. Median of time before the lesions were treated with platelets gel were 7 days. Lesions affected buccal mucosa, tongue, labial commissure and lower lip. Preliminar parameters were the microbiological contamination of lesions and presence of pain. Patients refer spontaneous widespread pain worsened by swallowing and feeding. Response to treatment has been evaluated in relation to the reduction of lesions dimensions, to the involution of pain and presence of granulation tissue after every application of platelet gel.

SUMMARY:
Oral mucositis (OM) is an inflammatory mucosal demolition frequently observed during treatments for neoplastic diseases such as chemotherapy or radiation therapy. The side effects of these treat-ments often drastically reduce patients' quality of life.

OM are the result of the systemic consequences of chemotherapy and radiotherapy which, due to their cytotoxic and local effects, lead to pain and severe ulceration with a consequent decrease in the quality of life of affected subjects. Plasma Rich in Fibrin is often used to enhance soft tissue wound healing and fight bacterial sepsis through the presence of leukocytes within it.

Aim of the retrospective study was to evaluate efficacy and safety of topic use of platelet gel in clinical management of oral mucositis in order to improve life quality of patients.

DETAILED DESCRIPTION:
Oral mucositis (OM) is a reversible common painful and debilitating iatrogenic lesion due to anti-cancer therapy. Depending on the intensity and dose of chemotherapy or radiotherapy, stomatitis or oral mucositis can significantly contribute to the reduction of patients' quality of life. [1]. The purpose of radiotherapy or chemotherapy therapies is to target rapidly duplicating cells and this triggers unwanted effects on oral and gastrointestinal mucosa, skin, bone marrow, hair follicles, and the tissues adjacent to the target [2].

OM can present with different characteristics of which the most common are edematous and ery-thematous areas, major ulcerations, pain and bleeding. In the most serious cases there is a diffi-culty in drinking, eating and speaking [3]. What is more, in severe cases it can damage patients' quality of life [4-5].

From a biochemical point of view, OM are caused by different molecular patterns such as oxida-tion produced by nitric oxide which causes cell apoptosis or the action of cyclooxygenases, protein kinases, cytokines and nuclear factors. Another interesting aspect to consider is the presence of epigenetic risk factors that target DNA methylation. [6,7] Oral mucositis mainly affects the non-keratinized oral mucosa as it has a cell turnover of 14 days which is twice as fast as keratinized gingiva. The areas of the oral cavity in which it is generally difficult to find this type of lesions are the hard palate, the dorsum of the tongue and the keratin-ized gingiva as they have a slower cell turnover (about 24 days) [8-9] To prevent the manifestation of these side effects, the guidelines of the Multinational Association of Supportive Care in Cancer and the International Society of Oral Oncology have defined home and professional oral hygiene as the main tool to combat OM, candidiasis and the risk of second-ary infections [10-15]. Care must be taken in removing all those mechanical traumas that can cause iatrogenic lesions such as incongruous margins, incongruous prostheses and grinding bites. However, it is also important to pay attention to all those external agents aggravating oral health such as tobacco, alcohol, oral burns and UV rays for the lips. Zinc supplements have also been suggested to maintain cellular homeostasis or human recombinant Keratinocyte Growth Factor to prevent oral mucositis. [13,16] OM lesions can also lead to large ulcers that can be terribly debilitating for patients. Scientific as-sociations for the protection of cancer patients recognize a key role in pain control and the prophy-laxis or treatment of secondary infections [12-15]. The use of low-intensity laser (Low-Level-Laser Therapy) was also proposed, which thanks to photobiostimulation can enhance tissue healing, re-duce inflammation and limit pain [12-15-17]. Zinc supplements are cofactors for many enzymes maintaining cellular equilibrium, immune response, and wound healing. They are considered an antioxidant, that precludes oxidative damage to many biomolecules [19]. In the most debilitating and painful cases of OM it has been suggested the use of a 2% morphine mouthwash and 0.5% doxepin mouthwash [13]. Furthermore, according to a study by O. Muhammad et al. [20], the glycyrrhetic acid / povidone / sodium hyaluronate gel could provide a mechanical protective action to the mucous membranes with a consequent reduction in pain.

Growth factors have been widely used in various fields of medicine and dentistry with the aim of improving and accelerating healing processes. The use of non-transfusional blood components such as Plasma Rich in Fibrin (PRF) is of great interest as it contains platelets and leukocytes can promote neoangiogenesis, release chemotactic growth factors and some studies have shown that leukocytes have a factor protective even in situations where there may be a risk of osteonecrosis. [21-22] Aim of the study is to evaluate efficacy and safety of topical use of platelet gel rich in fibrin in clinical management and healing of oral mucositis in oncological patients in treatment with chemotherapy and/or radiotherapy.

REFERENCIES:

1. Sroussi HY, Epstein JB, Bensadoun RJ, et al. Common oral complications of head and neck can-cer radiation therapy: mucositis, infections, saliva change, fibrosis, sensory dysfunctions, dental caries, periodontal disease, and osteoradionecrosis. Cancer Med 2017;6(12):2918-2931. DOI: 10.1002/cam4.122
2. White S, Pharoah M. Oral radiology: principles and interpretation, 7th ed. St. Louis: Elsevier; 2014
3. Bensinger W, Schubert M, Ang KK, Brizel D, Brown E, Eilers JG, et al. NCCN task force report. Prevention and management of mucositis in cancer care. J Natl Compr Canc Netw. 2008;6 Suppl 1:S1-21; quiz S22-24
4. Bensinger W, Schubert M, Ang KK, Brizel D, Brown E, Eilers JG, et al. NCCN task force report. Prevention and management of mucositis in cancer care. J Natl Compr Canc Netw. 2008;6 Suppl 1:S1-21; quiz S22-24
5. Baharvand M, Sarrafi M, Alavi K, Moghaddam EJ. Efficacy of topical phenytoin on chemothera-py-induced oral mucositis; a pilot study. Daru. 2010;18:46-50
6. Meyer-Hamme G, Beckmann K, Radtke J, Efferth T, Greten HJ, Rostock M, et al. A survey of chinese medicinal herbal treatment for chemotherapy-induced oral mucositis. Evid Based Com-plement Alternat Med. 2013;2013:284959
7. Carulli G, Rocco M, Panichi A, Chios CF, Ciurli E, Mannucci C, et al. Treatment of oral mucositis in hematologic patients undergoing autologous or allogeneic transplantation of peripheral blood stem cells: a prospective, randomized study with a mouthwash containing Camelia Sinensis leaf extract. Hematol Rep. 2013;5:21-25
8. Squier C, Brogden K. Human oral mucosa. Chichester, West Sussex, U.K.: Wiley-Blackwell; 2011
9. White S, Pharoah M. Oral radiology: principles and interpretation, 7th ed. St. Louis: Elsevier; 2014
10. Al-Ansari S, Zecha JAEM, Barasch A, de Lange J, Rozema FR, Raber- Durlacher JE. Oral mu-cositis induced by anticancer therapies. Curr Oral Health Rep (2015) 2:202-11. doi:10.1007/s40496-015-0069-4
11. Picardi A, Miranda M, Liciani F, Paterno G, Arcese W, Bollero P. Identification of oral risk fac-tors for chronic graft versus host disease in haematological patients who underwent allogeneic haematopoietic stem cell transplantation. Oral Implantol (Rome). 2017 Jan 21;10(4):390-397. doi:10.11138/orl/2017.10.4.390. eCollection 2017 Oct-Dec. PubMed PMID: 29682256;PubMed Cen-tral PMCID: PMC5892662.
12. Lalla RV, Sonis ST, Peterson DE. Management of oral mucositis in patients who have cancer. Dent Clin North Am (2008) 52(1):61-77,viii. doi:10.1016/j. cden.2007.10.002
13. Lalla RV, Bowen J, Barasch A, Elting L, Epstein J, Keefe DM, et al. MASCC/ ISOO clinical prac-tice guidelines for the management of mucositis secondary to cancer therapy. Cancer (2014) 120(10):1453-61. doi:10.1002/cncr.2859 14 Lalla RV. The MASCC/ISOO mucositis guidelines update: introduction to the first set of articles. Support Care Cancer (2013) 21(1):301-2. doi:10.1007/ s00520-012-1660-z

15) Lalla RV, Ashbury FD. The MASCC/ISOO mucositis guidelines: dissemination and clinical im-pact. Support Care Cancer (2013) 21(11):3161-3. doi:10.1007/s00520-013-1924-2 16) Bollero P., Franco R., Gianfreda F., Gualtieri P., Miranda M., Barlattani A. Epidemiology, Eti-opathogenesis, Treatment and Prognosis of Oral Thermal Burns from Food and Drinks. Dental Hy-potheses 2019. 10. 80. 10.4103/denthyp.denthyp_56_19.

17) Avci P, Gupta A, Sadasivam M, et al. Low-level laser (light) therapy (LLLT) in skin: stimulating, healing, restoring. Semin Cutan Med Surg 2013;32(1):41-52 18) Bollero, P., Rocco, F., Gianfreda, F., Miranda, M., Ottria, L., & Barlattani, A. (2019). The influ-ence of pemphigus vulgaris on oral health. ORAL & IMPLANTOLOGY, 12(2), 174-179.

19) Lin P, Sermersheim M, Li H, et al. Zinc in wound healing modulation. Nutrients 2017;10(1):E16. DOI: 10.3390/nu10010016 20) Maria OM, Eliopoulos N, Muanza T. Radiation-Induced Oral Mucositis. Front Oncol. 2017 May 22;7:89. doi: 10.3389/fonc.2017.00089 21) Picardi A, Ferraro AS, Miranda M, Meconi F, Lanti A, Adorno G, Arcese W, Bollero P. Therapeu-tic efficiency of platelet gel for the treatment of oral ulcers related to chronic graft versus host disease after allogeneic haematopoietic stem cell transplantation. Oral Implantol (Rome). 2017 Jan 21;10(4):398-405. doi: 10.11138/orl/2017.10.4.398. eCollection 2017 Oct-Dec. PubMed PMID: 29682257; PubMed Central PMCID: PMC5892654 22) Cantore S, Crincoli V, Boccaccio A, Uva AE, Fiorentino M, Monno G, Bollero P, Derla C, Fabiano F, Ballini A, Santacroce L. Recent Advances in Endocrine, Metabolic and Immune Disorders: Mes-enchymal Stem Cells (MSCs) and Engineered Scaffolds. Endocr Metab Immune Disord Drug Tar-gets. 2018;18(5):466-469. doi:10.2174/1871530318666180423102905. Review. PubMed PMID: 29692270.

ELIGIBILITY:
Inclusion Criteria:

All patients were affected by oral mucositis (9 RIOM, 6 chemotherapy-related oral mucositis). They were treated with almost 2 different systemic therapies before and during platelets gel applications. Median of time before the lesions were treated with platelets gel were 7 days. Lesions affected buccal mucosa, tongue, labial commissure and lower lip. Preliminar parameters were the microbiological contamination of lesions and presence of pain.

Exclusion Criteria:

Systemic Healthy Patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients were affected by oral mucositis due to RIOM or chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2021-07-19 (Actual)

PRIMARY OUTCOMES:
Complete Oral Mucositis Healing | 1 week
  Healing of oral lesions

CONTACTS AND LOCATIONS:
Overall Officials: Patrizio Bollero, Dentistry, Study Director — University of Rome Tor Vergata
Locations (1):
- Francesco Gianfreda, Taviano, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sroussi HY, Epstein JB, Bensadoun RJ, Saunders DP, Lalla RV, Migliorati CA, Heaivilin N, Zumsteg ZS. Common oral complications of head and neck cancer radiation therapy: mucositis, infections, saliva change, fibrosis, sensory dysfunctions, dental caries, periodontal disease, and osteoradionecrosis. Cancer Med. 2017 Dec;6(12):2918-2931. doi: 10.1002/cam4.1221. Epub 2017 Oct 25. PMID 29071801
- [Background] Bensinger W, Schubert M, Ang KK, Brizel D, Brown E, Eilers JG, Elting L, Mittal BB, Schattner MA, Spielberger R, Treister NS, Trotti AM 3rd. NCCN Task Force Report. prevention and management of mucositis in cancer care. J Natl Compr Canc Netw. 2008 Jan;6 Suppl 1:S1-21; quiz S22-4. PMID 18289497
- [Background] Agren MS, Rasmussen K, Pakkenberg B, Jorgensen B. Growth factor and proteinase profile of Vivostat(R) platelet-rich fibrin linked to tissue repair. Vox Sang. 2014 Jul;107(1):37-43. doi: 10.1111/vox.12120. Epub 2013 Dec 10. PMID 24320875
- [Background] Hirase T, Ruff E, Surani S, Ratnani I. Topical application of platelet-rich plasma for diabetic foot ulcers: A systematic review. World J Diabetes. 2018 Oct 15;9(10):172-179. doi: 10.4239/wjd.v9.i10.172. PMID 30364787